CLINICAL TRIAL: NCT02158923
Title: Postoperative Complication and Hospital Stay Reduction With a Individualized Perioperative Lung Protective Ventilation. A Comparative, Prospective, Multicenter, Randomized Controlled Trial.
Brief Title: Individualized Perioperative Open Lung Ventilatory Strategy
Acronym: iPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Hospital de Manises (Other); Hospital General Valencia (Other); Hospital Universitario La Fe (Other); Germans Trias i Pujol Hospital (Other); Hospital de Sant Pau (Other); Hospital del Mar (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital General Universitario de Alicante (Other); Hospital Juan Canalejo (Other); Hospital General Regional de León (Other Government); Hospital Universitario Virgen de la Arrixaca (Other); Hospital Miguel Servet (Other); Hospital Clínico Universitario de Valladolid (Other); Hospital Universitario Fundación Alcorcón (Other); Hospital General de Ciudad Real (Other); Hospital Universitario de Valme (Other); Hospital de Basurto (Other); Hospital Dr. Negrín (Unknown); Hospital de Galdakano (Unknown); Complejo Hospitalario de Especialidades Juan Ramón Jimenez (Other); Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Carlos Ferrando, MD, PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: iPROVE
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Moderated-high Risk of Postoperative Pulmonary Complication; Abdominal Surgery Expected More Than Two Hours
Keywords: ventilation; lung; lung complications; postoperative complications; perioperative lung protective ventilation
MeSH Terms: conditions — Respiratory Aspiration; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Individualized ventilation (Experimental): Intraoperatively ventilated patients with a tidal volume (VT) of 8 ml / kg of ideal body weight, and a FiO2 of 0.8. After intubation, all patients were conduct an alveolar recruitment maneuver (MRA) and PEEP level individualized spanned (see Calculation of optimal PEEP). Every 40 minutes will be assessed the need to adjust the level of PEEP by evaluating the dynamic compliance of the respiratory system (Crs). Faced with a decline in Crs> 10% a new MRA and optimal PEEP setting will be assessed.
  Interventions: Procedure: Alveolar recruitment maneuver; Procedure: Calculation of optimal PEEP
- Individualized vent. + postop. CPAP (Experimental): Intraoperatively ventilated patients with a tidal volume of 8 ml / kg of ideal body weight, and a FiO2 of 0.8. After intubation, all patients were conduct an alveolar recruitment maneuver (MRA) and PEEP level individualized spanned (see Calculation of optimal PEEP). Every 40 minutes will be assessed the need to adjust the level of PEEP by evaluating the dynamic compliance of the respiratory system (Crs). Faced with a decline in Crs> 10% a new MRA and optimal PEEP setting will be assessed. Postoperatively a CPAP of 5 cmH2O (or 10 cmH2O if BMI> 30) with a FiO2 of 0.5 will be applied.
  Interventions: Procedure: Alveolar recruitment maneuver; Procedure: Calculation of optimal PEEP; Procedure: Postoperative CPAP
- Standard ventilation (No Intervention): Intraoperatively ventilated patients with a tidal volume of 8 ml / kg of ideal body weight, PEEP 6 cmH2O and FiO2 0.8. In these groups no recruitment maneuvers or optimal PEEP setting will be performed.
- Standard vent. + postoperative CPAP (Active Comparator): Intraoperatively ventilated patients with a tidal volume of 8 ml / kg of ideal body weight, PEEP 6 cmH2O and FiO2 0.8. In these groups no recruitment maneuvers or optimal PEEP setting will be performed. Postoperatively, a CPAP of 5 cmH2O (or 10 cmH2O if BMI> 30) with a FiO2 of 0.5 will be applied.
  Interventions: Procedure: Postoperative CPAP

INTERVENTIONS:
Procedure: Alveolar recruitment maneuver — To start Alveolar Recruitment Maneuver (ARM), change ventilatory pressure-controlled mode (PCV) with 15 cmH2O pressure control ventilation. A respiratory rate (RR) of 15 rpm, inspiration: expiration ratio of 1:1, FiO2 of 0.8 and PEEP of 10 cmH2O. PEEP level will increase 5 on 5 cmH2O every 10 respiratory cycles, increasing to 15 cycles in the last level of PEEP (25 cmH2O), getting an opening pressure at 40 cmH2O airway (duration of the maneuver: 160 sec.)
  Arms: Individualized vent. + postop. CPAP; Individualized ventilation
Procedure: Calculation of optimal PEEP — Change ventilation mode to volume controlled ventilation (VCV) with a VT of 8 ml / kg, RR 15 rpm and adjust a PEEP of 20 cmH2O. Descend PEEP level 2 by 2 cmH2O every 30 seconds until obtain the best respiratory system compliance (Crs) PEEP. Once you know the optimal level of PEEP (best Crs PEEP), will be conducted again alveolar recruitment maneuver and adjust the best Crs level of PEEP + 2 cmH2O .
  Arms: Individualized vent. + postop. CPAP; Individualized ventilation
Procedure: Postoperative CPAP — Postoperatively, non-invasive mechanical ventilation with a CPAP of 5 cmH2O (or 10 cmH2O if BMI> 30) with a FiO2 of 0.5 will be applied.
  Arms: Individualized vent. + postop. CPAP; Standard vent. + postoperative CPAP

SUMMARY:
The purpose of this study is to determine whether individualized ventilatory management combining the use of low tidal volumes, alveolar recruitment maneuvers, individually titrated positive end-expiratory pressure and postoperative individualized ventilatory support will decrease postoperative complications, unplanned ICU readmissions, ICU and hospital length of stay and mortality compared to a standardized Lung Protective Ventilation (LPV) for all patients at risk.

ELIGIBILITY:
Inclusion Criteria:

* Age not less than 18
* Risk of postoperative pulmonary complication moderate-high defined by a score ≥ 26 on the risk scale ARISCAT (based on the analysis of seven factors, where a score between 26 and 44 points defines a moderate risk, and a score> 44 points define a high risk, included in the Information Booklet Investigator).
* Planned abdominal surgery> 2 hours.
* Signed informed consent for participation in the study.

Exclusion Criteria:

* Age less than 18 years.
* Pregnant or breast-feeding.
* Patients with BMI >35.
* Syndrome of moderate or severe respiratory distress: PaO2/FiO2 < 200 mmHg.
* Heart failure: NYHA IV.
* Hemodynamic failure: CI <2.5 L/min/m2 and / or requirements before surgery ionotropic support.
* Diagnosis or suspicion of intracranial hypertension (intracranial pressure> 15 mmHg).
* Mechanical ventilation in the last 15 days.
* Presence of pneumothorax. Presence of giant bullae on chest radiography or computed tomography (CT).
* Patient with preoperatively CPAP.
* Participation in another experimental protocol at the time of intervention selection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Reduction of lung and systemic postoperative complications | Up to 7 postoperative days

SECONDARY OUTCOMES:
Reduction of lung and systemic postoperative complications | Up to 30 postoperative days

OTHER OUTCOMES:
Mortality evaluation | 180 and 365 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ferrando, MD, PhD, Study Director — Hospital Clínico Universitario Valencia
Locations (7):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Hospital Privado de la Comunidad, Mar del Plata, Buenos Aires, Argentina
- Spain (4):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Department of Anesthesia and Critical Care; Hospital Clinico Universitario, Valencia, Valencia
- Uppsala University Hospital, Uppsala, Uppland, Sweden

REFERENCES:
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] PROVE Network Investigators for the Clinical Trial Network of the European Society of Anaesthesiology; Hemmes SN, Gama de Abreu M, Pelosi P, Schultz MJ. High versus low positive end-expiratory pressure during general anaesthesia for open abdominal surgery (PROVHILO trial): a multicentre randomised controlled trial. Lancet. 2014 Aug 9;384(9942):495-503. doi: 10.1016/S0140-6736(14)60416-5. Epub 2014 Jun 2. PMID 24894577
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Derived] Ferrando C, Librero J, Tusman G, Serpa-Neto A, Villar J, Belda FJ, Costa E, Amato MBP, Suarez-Sipmann F; iPROVE Network Group. Intraoperative open lung condition and postoperative pulmonary complications. A secondary analysis of iPROVE and iPROVE-O2 trials. Acta Anaesthesiol Scand. 2022 Jan;66(1):30-39. doi: 10.1111/aas.13979. Epub 2021 Sep 22. PMID 34460936
- [Derived] Garutti I, Errando CL, Mazzinari G, Bellon JM, Diaz-Cambronero O, Ferrando C; iPROVE network. Spontaneous recovery of neuromuscular blockade is an independent risk factor for postoperative pulmonary complications after abdominal surgery: A secondary analysis. Eur J Anaesthesiol. 2020 Mar;37(3):203-211. doi: 10.1097/EJA.0000000000001128. PMID 32028288
- [Derived] Ferrando C, Soro M, Unzueta C, Suarez-Sipmann F, Canet J, Librero J, Pozo N, Peiro S, Llombart A, Leon I, India I, Aldecoa C, Diaz-Cambronero O, Pestana D, Redondo FJ, Garutti I, Balust J, Garcia JI, Ibanez M, Granell M, Rodriguez A, Gallego L, de la Matta M, Gonzalez R, Brunelli A, Garcia J, Rovira L, Barrios F, Torres V, Hernandez S, Gracia E, Gine M, Garcia M, Garcia N, Miguel L, Sanchez S, Pineiro P, Pujol R, Garcia-Del-Valle S, Valdivia J, Hernandez MJ, Padron O, Colas A, Puig J, Azparren G, Tusman G, Villar J, Belda J; Individualized PeRioperative Open-lung VEntilation (iPROVE) Network. Individualised perioperative open-lung approach versus standard protective ventilation in abdominal surgery (iPROVE): a randomised controlled trial. Lancet Respir Med. 2018 Mar;6(3):193-203. doi: 10.1016/S2213-2600(18)30024-9. Epub 2018 Jan 19. PMID 29371130
- [Derived] Ferrando C, Soro M, Canet J, Unzueta MC, Suarez F, Librero J, Peiro S, Llombart A, Delgado C, Leon I, Rovira L, Ramasco F, Granell M, Aldecoa C, Diaz O, Balust J, Garutti I, de la Matta M, Pensado A, Gonzalez R, Duran ME, Gallego L, Del Valle SG, Redondo FJ, Diaz P, Pestana D, Rodriguez A, Aguirre J, Garcia JM, Garcia J, Espinosa E, Charco P, Navarro J, Rodriguez C, Tusman G, Belda FJ; iPROVE investigators (Appendices 1 and 2). Rationale and study design for an individualized perioperative open lung ventilatory strategy (iPROVE): study protocol for a randomized controlled trial. Trials. 2015 Apr 27;16:193. doi: 10.1186/s13063-015-0694-1. PMID 25927183